CLINICAL TRIAL: NCT01751841
Title: Outcome Analysis for Minimally Invasive Spine Surgery and Navigation
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 19-12021199
Record Dates: First submitted 2012-11-07; First posted 2012-12-18 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal fusion patients with minimally invasive spine surgery: Spinal fusion patients for whom Silicate-Substituted Calcium Phosphate Ceramic has been used as the Bone Graft

SUMMARY:
Prospective/Retrospective data analysis, chart reviews and clinical outcomes of minimally invasive spine surgery

DETAILED DESCRIPTION:
STUDY RATIONALE AND PRIMARY OBJECTIVE/HYPOTHESIS To assess the clinical and radiographic outcome of spinal fusion procedures using Silicate-Substituted Calcium Phosphate (Si-CaP), a newer-generation of synthetic ceramics designed to maximize osteoinduction and osteoconduction.

STUDY DESIGN Retrospective Study

PURPOSE OF THE STUDY Providing compelling evidence for the efficacy of Si-CaP in terms of resulting in satisfactory fusion.

SUMMARY OF METHODS A prospectively collected database will be reviewed retrospectively, to retrieve data of 200 patients who have undergone different spinal fusion procedures using Silicate-Substituted Calcium Phosphate (Si-CaP). An average follow up duration of at least 12 months will be considered. Clinical outcomes will be assessed using the visual analog scale (VAS), Oswestry Disability Index (ODI), and Neck Disability Index (NDI). Pre-operative scores will be compared to the latest follow-up scores. A board certified Neuro-radiologist will assess the fusion rate. Fusion will be determined by the presence of bony bridging on 2 consecutive sections in at least 2 planes on computed tomographic imaging.

SECONDARY ENDPOINTS AND EXPECTED RESULTS The purpose of this study is to evaluate the level of clinical and radiographic improvement in patients implanted with Silicate-Substituted Calcium Phosphate (Si-CaP) as a bone graft substitute material for spinal fusions. More comprehensive long term studies will be able to provide compelling evidence for the efficacy of Si-CaP in terms of resulting in satisfactory fusion. They can more strongly support the previously published data implying that Si-CaP can be utilized as an alternative to autogenous bone graft in spinal arthrodesis procedures.

ELIGIBILITY:
Inclusion Criteria:

- Patients with different spinal fusion procedures (including axial lumbar interbody fusion, transforaminal lumbar interbody fusion, extreme lateral interbody fusion, posterior cervical fusion, and anterior discectomy and fusion using Silicate-Substituted Calcium Phosphate as a bone graft substitute.

Exclusion Criteria:

- Utilization of any other bone extenders in addition to Si-CaP as a bone graft substitute.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our prospectively collected institutional database will be reviewed to identify all consecutive patients with spinal fusion procedures using Silicate-Substituted Calcium Phosphate as a bone graft substitute. Surgeries have been performed at our hospital between 2007 and 2011. The estimated number of patients enrolled in the study is 200 patients. Patient demographics will be extracted using the database. The study population are from different age, gender and ethnicity groups. The indications for surgery will be recorded for each patient, as well. Institutional Research Board approval has been granted. All patients have provided informed consent for data collection regarding their treatment and outcomes.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Up to 2 years
  Pre-operative pain scores will be compared to the latest follow-up pain scores.

SECONDARY OUTCOMES:
Fusion on CT imaging or flexion-extension radiographs. | Up to 2 years
  A board certified Neuro-radiologist will assess the fusion rate.Fusion will be determined by the presence of bony bridging on 2 consecutive sections in at least 2 planes on computed tomographic imaging.
Oswestry Disability Index (ODI) | Up to 2 years
  Pre-operative scores will be compared to the latest follow-up scores.
Neck Disability Index (NDI) | Up to 2 years
  Pre-operative scores will be compared to the latest follow-up scores.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Härtl, MD, Principal Investigator — Weill Cornell Neurological Surgery Department
Locations (1):
- Weill Cornell Brain and Spine Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nagineni VV, James AR, Alimi M, Hofstetter C, Shin BJ, Njoku I Jr, Tsiouris AJ, Hartl R. Silicate-substituted calcium phosphate ceramic bone graft replacement for spinal fusion procedures. Spine (Phila Pa 1976). 2012 Sep 15;37(20):E1264-72. doi: 10.1097/BRS.0b013e318265e22e. PMID 22744618
- See also: Silicate-substituted calcium phosphate ceramic bone graft replacement for spinal fusion procedures. — http://www.ncbi.nlm.nih.gov/pubmed/22744618